CLINICAL TRIAL: NCT00000825
Title: A Randomized, Open-Label Phase II Study of Subcutaneous Interleukin-2 (Proleukin) Plus Antiretroviral Therapy vs. Antiretroviral Therapy Alone in Patients With HIV Infection and at Least 350 CD4+ Cells/mm3
Brief Title: The Effects of Giving Interleukin-2 (IL-2) Plus Anti-HIV Therapy to HIV-Positive Patients With CD4 Cell Counts of at Least 350 Cells/mm3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: IRP 021C; 10466 (Registry Identifier: DAIDS ES); SQIL-2; SQIL-2 Houston
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV-1; Interleukin-2; Dose-Response Relationship, Drug; Antiviral Agents; CD4 Lymphocyte Count; DNA, Viral
MeSH Terms: conditions — HIV Infections | interventions — aldesleukin

INTERVENTIONS:
Drug: Aldesleukin

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of giving IL-2 plus anti-HIV (antiretroviral) therapy to HIV-positive patients with CD4 cell counts (cells of the immune system that fight infection) of at least 350 cells/mm3. This study will also examine the ability of antiretroviral therapy combined with IL-2 to boost the immune system.

IL-2, given through injection under the skin, in combination with anti-HIV therapy can increase CD4 cell counts. This study examines 3 doses of IL-2 in order to determine the safest and most effective dose to use.

DETAILED DESCRIPTION:
IL-2, administered subcutaneously in combination with antiretrovirals, has resulted in increased CD4+ cell counts which may retard HIV disease progression. Using a smaller patient sampling, this Phase II study helps develop the clinical experience needed to consider formation of a larger, more complete Phase III trial.

Seventy-two HIV-infected patients (previously treated or naive) are randomized independently to receive either control therapy with antiretrovirals alone OR escalating doses of subcutaneous interleukin-2 (IL-2) plus antiretrovirals. In the absence of dose-limiting toxicity (DLT) in at least 9 of 12 patients in Group 1, 12 additional patients are entered into Group 2 and treated as indicated. In the absence of DLT in 9 of 12 patients in Group 2, the final 12 patients are entered into Group 3. Those patients enrolled in either of the first 2 dose groups who complete 3 courses of therapy have their dose escalated to a maximum dose. A course of treatment is defined as 5 days of IL-2 plus antiretrovirals followed by 7 weeks of antiretroviral therapy alone.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Have a CD4 cell count greater than or equal to 300 cells/mm3.
* Have no AIDS-defining illnesses.
* Are at least 18 years old.
* Have been on antiretroviral therapy for at least 7 days prior to study entry.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Abuse alcohol or drugs, or have any serious psychiatric or medical illnesses that would affect their safety or ability to complete the study.
* Have a history of the following: cancer (other than Kaposi's sarcoma), an AIDS-defining illness, a central nervous system abnormality, or an autoimmune/inflammatory disease.
* Are pregnant or breast-feeding.
* Have ever received IL-2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72
Dates: Start 1998-05; Primary Completion 2000-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Street Clinic C605-020 CRS, Houston, Texas, United States